CLINICAL TRIAL: NCT05382884
Title: The SUPPORT Study: Survey and Development of a Universally Accessible Postpartum Online Resource for the Treatment of Postpartum Depression
Brief Title: The SUPPORT Study: Effectiveness and Usability of a Web-Enabled Resource for Postpartum Mental Health
Acronym: SUPPORT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Women's Health Research Institute of British Columbia (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Lori Brotto, Director, UBC Sexual Health Laboratory, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H21-03407
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-05

CONDITIONS: Postpartum Depression; Postpartum Anxiety; Postnatal Depression; Perinatal Disorder; Perinatal Depression; Postpartum Disorder
Keywords: Postpartum Depression; Postpartum Anxiety; Perinatal; Postnatal; eHealth; Online Intervention; Website; Web-Enabled
MeSH Terms: conditions — Depression, Postpartum; Puerperal Disorders

STUDY DESIGN:
Intervention Model Description: The present study phase uses a randomized controlled trial design and will evaluate the effectiveness and usability of postpartumcare.ca. Fifty participants will be randomized to the intervention group, receiving immediate access to postpartumcare.ca for 4 weeks, and 50 will be assigned to a waitlist control group, receiving treatment as usual for the duration of the 4-week intervention period. Following the 4-week intervention period and 2-week follow-up, participants from both groups will be able to access postpartumcare.ca.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Fifty participants will be randomized to the intervention group, receiving immediate access to postpartumcare.ca for a period of 4 weeks. Intervention group participants may use postpartumcare.ca as often as desired for the duration of the 4-week intervention period. Following the 4-week intervention period and a 2-week follow-up period, intervention group participants will retain access to postpartumcare.ca.
  Interventions: Other: Postpartumcare.ca (Web-Enabled Intervention)
- Waitlist Control (No Intervention): Fifty participants will be randomized to a waitlist control group, receiving treatment as usual (TAU) for a period of 4 weeks. Following the 4-week intervention period and a 2-week follow-up period, waitlist control participants will receive access to postpartumcare.ca.

INTERVENTIONS:
Other: Postpartumcare.ca (Web-Enabled Intervention) — Postpartumcare.ca is a web-enabled intervention accessible via computer, tablet or smartphone devices. The content and design of postpartumcare.ca were created based on the needs, opinions, and desires of birthing parents in British Columbia affected by postpartum depression and/or anxiety, which were solicited previously in phases 1 & 2 of the SUPPORT study.
  Arms: Intervention

SUMMARY:
The SUPPORT Study aims to evaluate the effectiveness and usability of postpartumcare.ca, a web-enabled resource for postpartum depression (PPD) and postpartum anxiety (PPA), created based on the input of birthing parents in British Columbia (BC) affected by these disorders.

DETAILED DESCRIPTION:
This is Phase 3 of a multi-phase project that will be completed under the supervision of Dr. Lori Brotto, the University of British Columbia Sexual Health Lab and the Women's Health Research Institute at BC Women's Hospital.

The present study phase uses a randomized controlled trial design and will evaluate the effectiveness and usability of postpartumcare.ca using three outcomes: (1) depression and anxiety; (2) system usability and satisfaction; and (3) website metrics. Parents aged 19 or older experiencing postpartum depression and/or anxiety living in BC who gave birth in the past 12 months will be eligible. Fifty will be randomized to the intervention group, receiving immediate access to postpartumcare.ca for 4 weeks, and 50 will be assigned waitlist control, receiving treatment as usual.

Depression and anxiety symptoms will be measured at baseline, after the 4-week intervention period, and again 2 weeks later using the Edinburgh Postnatal Depression Scale (EPDS) and Perinatal Anxiety Screening Scale (PASS). After 4 weeks, system usability and satisfaction will be measured using the System Usability Scale (SUS), and website metrics will be collected for the intervention group only.

Multivariate analyses will be conducted to compare the anxiety and depression total scores and subscale scores between the two groups (intervention and treatment as usual). Descriptive analyses will be conducted on the satisfaction and usability questionnaires and website metrics.

The investigators hypothesize that following the use of postpartumcare.ca, the intervention group will see a greater reduction in depression and/or anxiety symptoms compared to the control group and that the website will be rated as usable.

The findings from this trial will add to the existing body of literature investigating the use of eHealth interventions for PPD and PPA treatment. Moreover, postpartumcare.ca will serve as a practical tool for birthing persons in BC in need of accessible and effective support.

ELIGIBILITY:
Inclusion Criteria:

* have given birth within the past 12 months
* reside in British Columbia
* be at least 19 years of age
* have the ability to communicate in English
* have a suspected diagnosis or symptoms of postpartum depression and/or anxiety, as measured by the Edinburgh Depression Scale, having a score of 9 or greater and/or PASS score of 26 or greater, as measured as part of the initial eligibility questionnaire
* have access to study materials online, that is, have internet access and a device to access the internet, such as a computer or smartphone

Exclusion Criteria:

* have not given birth within the past 12 months
* reside outside of British Columbia
* under 19 years of age
* unable to communicate in English
* do not have a suspected diagnosis or symptoms of postpartum depression and/or anxiety, as measured by the Edinburgh Depression Scale, having a score of 8 or less and/or PASS score of 25 or less, as measured as part of the initial eligibility questionnaire
* do not have any internet access

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Postpartum Depression at 4 weeks and 6 weeks, evaluated using the Edinburgh Postnatal Depression Scale (EPDS). | The EPDS will be administered at baseline, after a 4-week intervention period, and again after a 2-week follow up period
  Changes in postpartum depression will be evaluated using the Edinburgh Postnatal Depression Scale (EPDS). The EPDS is a standard scale used internationally to evaluate postpartum depression in the clinical setting and is recommended for screening of all postpartum parents who gave birth in British Columbia. Scoring on the EPDS ranges from 0 to 30, with higher scores indicating more severe depressive symptoms.
Change from Baseline Postpartum Anxiety at 4 weeks and 6 weeks, evaluated using the Perinatal Anxiety Screening Scale (PASS). | The PASS will be administered at baseline, after a 4-week intervention period, and again after a 2-week follow up period
  Changes in postpartum anxiety will be evaluated using the Perinatal Anxiety Screening Scale (PASS). The PASS is a commonly used measure for screening for anxiety in the perinatal period. Scoring on the PASS ranges from 0 to 93, with higher scores indicating more severe anxiety symptoms
Website usability, as evaluated using the System Usability Scale (SUS) | Website usability will be evaluated after the 4-week intervention period for the intervention group only
  Usability of the website intervention will be measured using a modified version of the System Usability Scale (SUS). The SUS is a reliable tool for measuring usability consisting of a 10-item questionnaire with 5 response options ranging from Strongly Agree to Strongly Disagree.
Website satisfaction, evaluated using the Patient Global Impression of Change (PGIC) questionnaire | Website satisfaction will be evaluated after the 4-week intervention period for the intervention group only
  Satisfaction with the website intervention will be measured using a brief Patient Global Impression of Change (PGIC) questionnaire developed for this study. the PGIC describes a participant's belief about the efficacy of treatment on a 7 point scale where change is rated as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse.".
Website satisfaction, evaluated using the user-perceived web quality instrument | Website satisfaction will be evaluated after the 4-week intervention period for the intervention group only
  Satisfaction with the website intervention will be measured using the user-perceived web quality instrument. The user perceived web quality instrument is a 25-item instrument that measures four dimensions of web quality: specific content, content quality, appearance and technical adequacy.
Website satisfaction, evaluated using the Patient Education Materials Assessment Tool (PEMAT) | Website satisfaction will be evaluated after the 4-week intervention period for the intervention group only
  Satisfaction with the website intervention will be measured using the Patient Materials Assessment Tool (PEMAT). The PEMAT evaluates and compares the understandability and actionability of patient education materials using a 26-item scale.
Website metrics including average time on page, average session duration, returning visitors, and number of pages visited per session. | Website metrics will be collected after the 4-week intervention period for the intervention group only
  Website metrics describe how participants use the website intervention. Included website metrics will be average time on page, average session duration, returning visitors, and the number of pages visited per session. These metrics will be collected using Matomo Analytics.

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Heath Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lawrence CG, Breau G, Yang L, Hellerstein OS, Hippman C, Kennedy AL, Ryan D, Shulman B, Brotto LA. Effectiveness of a web-enabled psychoeducational resource for postpartum depression and anxiety among women in British Columbia. Arch Womens Ment Health. 2024 Dec;27(6):995-1010. doi: 10.1007/s00737-024-01468-8. Epub 2024 May 6. PMID 38709329